CLINICAL TRIAL: NCT02048137
Title: Transcranial Direct Current Stimulation to Reduce Chronic Pain in Patients With Chronic Inflammatory Bowel Diseases
Acronym: tDCS in IBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Magdalena S. Prüß née Volz, Dr. med. Magdalena Volz, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA4/135/13; EA4/135/13 (Other: Charité Universitätsmedizin Berlin)
Record Dates: First submitted 2014-01-11; First posted 2014-01-29 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active transcranial direct current stimulation (Active Comparator)
  Interventions: Device: Transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation

SUMMARY:
In the study we test whether transcranial direct current stimulation can reduce the perception of pain in patients with chronic inflammatory bowel diseases.

Hypothesis: Transcranial direct current stimulation can reduce the perception of pain in patients with chronic inflammatory bowel diseases.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease
* Chronic pain (more than 3 months)
* Pain (VAS > 3/10)

Exclusion Criteria:

* Contraindication to transcranial direct current stimulation
* Pregnancy
* Sever internal or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | 1 week

SECONDARY OUTCOMES:
Visual analoug scale - pain | 1 week

OTHER OUTCOMES:
Quality of life | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University Medicine, Berlin, Germany

REFERENCES:
- See also: Related Info — http://gastro.charite.de/en/
- See also: Department of Gastroenterology, Infectiology and Rheumatology (including workspace nutrition medicine) — http://gastro.charite.de/en/